CLINICAL TRIAL: NCT03719404
Title: Effect of Irrigants on Outcome of Non Surgical Endodontic Retreatment: A Randomised Controlled Trial
Brief Title: Irrigants on Outcome of Non Surgical Endodontic Retreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Kaarunya
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Root Canal Infection
Keywords: Retreatment; Irrigants; chlorhexidine
MeSH Terms: interventions — Sodium Hypochlorite; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sodium hypochlorite group (Experimental): sodium hypochlorite and EDTA are used in endodontic retreatment cases
  Interventions: Procedure: sodium hypochlorite
- chlorhexidine group (Experimental): chlorhexidine and citric acid are used in endodontic retreatment cases
  Interventions: Procedure: chlorhexidine

INTERVENTIONS:
Procedure: sodium hypochlorite — sodium hypochlorite is used as primary irrigant and edta is used as secondary irrigant in endodontic retreatment cases
  Arms: sodium hypochlorite group
Procedure: chlorhexidine — Chlorhexidine is used as primary irrigant and citric acid is used as secondary irrigant in endodontic retreatment cases
  Arms: chlorhexidine group

SUMMARY:
Till date, no study has systematically evaluated the role of a single variable on success of endodontic retreatment. While the evaluation of a single factor as the primary objective in a study is a difficult task, it unarguably provides more valuable information regarding the influence of that variable on outcome. The clinical studies comparing the use of Sodium hypochlorite (NaOCl) and Chlorhexidine digluconate (CHX) in retreatment cases have evaluated only the antibacterial effectiveness and there is no clinical study comparing their effect on the clinical outcome in retreatment cases. And also, no study has compared the use of irrigant as single variable in the primary objective on success of retreatment cases. The conclusions drawn from such "surrogate measures" must be interpreted and applied in clinical settings with caution. Since there is no standardised irrigation treatment protocol for secondary root canal treatment, the present study is being conducted to evaluate the effect of 5% NaOCl with 17% Ethylenediaminetetraacetic acid (EDTA) and 2% CHX with 10% citric acid (CA) on outcome, when used as irrigants during the chemomechanical preparation in retreatment cases.

DETAILED DESCRIPTION:
Introduction: Retreatment is defined as a procedure to remove root canal filling materials from the tooth, followed by cleaning, shaping and obturating the canals (AAE glossary of endodontic terms). There is a scarcity in retreatment studies when compared to literature available pertaining to primary root canal treatment. Till date, only 7 studies are available which have attempted to analyse the factors predicting the prognosis of nonsurgical retreatment. However, none of these studies has systematically evaluated the role of a single variable on success of endodontic retreatment. These are either retrospective or cohort studies, with no study identifiable as a randomised controlled trial. While the evaluation of a single factor as the primary objective in a study is a difficult task, it unarguably provides more valuable information regarding the influence of that variable on outcome. The present study is being conducted to evaluate the effect of 5% NaOCl with 17% EDTA, and 2% CHX with 10% CA on outcome, when used as irrigants during the chemomechanical preparation in retreatment cases.

Aim and Objectives: To evaluate and compare the success of nonsurgical endodontic retreatment following use of the two different irrigant regimes, using 5% NaOCl with 17% EDTA and 2% CHX with 10% CA.

Setting: Study subjects will be recruited from Post Graduate Department of Conservative Dentistry and Endodontics, PGIDS, Rohtak, Haryana.

Study design: Prospective randomized controlled trial Time frame: 18 months Method: Patients with above inclusion criteria will be selected and randomly allocated to one of the two study groups according to the irrigants used ( NaOCl + EDTA , CHX + CA ). The secondary root canal treatment was completed in two visits. Proper rubber dam isolation and aseptic conditions were followed throughout the procedure. Caries and /or coronal restorations were removed with sterile burs. The coronal two thirds of the root filling was mechanically removed with hand files. A sterile #15 K- file was used to create space by applying a gentle filing motion. A larger endodontic file was used to engage the root canal filling material and the file with the attached root filling material was withdrawn from the canal. The working length was determined with the aid of the electronic apex locator and radiographs using digital sensor (Carestream RVG 5200, Carestream Health Inc, Rochester, NY). Apical preparation was completed to the working length with hand stainless-steel files. 2 ml of corresponding chosen primary irrigant (NaOCl or CHX) was used after each instrument change in the respective groups. All the irrigation procedures were performed using a 30 gauge needle ensuring that the needle was placed to within 1-2mm from the apex. After preparation of the canals, the smear layer was removed using a rinse of 5 ml of either 17% EDTA or 10 % CA depending on the group, which was ultrasonically activated for 3 minutes. Then the final irrigation was done using 5 ml of corresponding primary irrigant of the group. The root canal walls were then dried using paper points. Calcium hydroxide paste mixed with sterile saline was placed with Lentulo spiral fillers in the entire root canal extent and the access cavity was restored with Cavit. The dressing was left in place for 7 days. At the second visit, the temporary restoration was removed. The intracanal dressing was removed with 5 ml of corresponding primary irrigant and with gentle filing with the use of Hedstroem file. The root canal was then irrigated with 5 ml of corresponding chelating agent with ultrasonic activation followed by 5 ml of primary irrigants of the corresponding group. The canals were dried and obturated with the GuttaPercha using lateral condensation technique and Zinc Oxide- Eugenol based sealer in both the groups. After obturation, the tooth was restored permanently. Immediate post-operative radiograph was then taken using preset exposure parameters with Rinn paralleling device. Follow up clinical and radiographic examinations were carried out every 3 months, till 12 months period.

Statistical analysis: The data gathered will be analyzed using suitable statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Previously root filled Permanent teeth with post-treatment apical periodontitis requiring nonsurgical root canal retreatment with clinical symptoms like pain on palpation and discomfort to percussion
* Radiographic evidence of periapical radiolucency (minimum size ≥ 2.0 × 2.0 mm)
* previous initial endodontic treatment was done atleast 4 years before.
* Patient's age more than 18 years.
* Patient willingness to participate in the study

Exclusion Criteria:

periodontal deep pockets more than 4mm, previous procedural errors, not suitable for rubber dam isolation, vertical root fractures, intraradicular post, marginal or furcal bone loss due to periodontitis, nonrestorable teeth and patients with diabetes, pregnancy, antibiotic medication within last three months, any systemic or immunocompromising conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Radiographic success | Baseline to one year
  Follow up will be done every 3 months till 12 months. Scoring of each tooth will be done according to the following five point scale (PAI). 1- normal periapical structures 2-Small changes in bone structure 3-Changes in bone structure with some mineral loss 4-Periodontitis with well-defined radiolucent area 5-Severe periodontitis with exacerbating features
  Instructions for scoring using PAI:
  * All teeth must be given a score
  * When in doubt assign higher score
  * For multirooted teeth, use the highest of the scores given to the individual roots.
  Success was calculated as a dichotomous variable with teeth showing a PAI score of ≤ 2 considered as healed, while those showing a score of ≥3 considered as nonhealed.

IPD SHARING:
Plan to Share IPD: No